CLINICAL TRIAL: NCT04285749
Title: Prevention of Recurrence and Metastasis in Genetically High-Risk Melanomas
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: PI moving to new institution prior to study activation
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE4619
Record Dates: First submitted 2020-02-24; First posted 2020-02-26 (Actual); Last update posted 2020-07-27 (Actual); Status verified 2020-07

CONDITIONS: Malignant Melanoma
MeSH Terms: conditions — Melanoma | interventions — Fluvastatin; Base Sequence; Gene Expression Profiling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Fluvastatin (Experimental): Participants will receive Fluvastatin for 2 weeks.
  RNA-sequencing and gene expression profiling will be completed on the original diagnostic biopsy and the final melanoma excision.
  Interventions: Drug: Fluvastatin; Other: RNA-sequencing; Other: Gene expression profiling

INTERVENTIONS:
Drug: Fluvastatin — Fluvastatin PO 80mg QD for 2 weeks
Other: RNA-sequencing — RNA-sequencing will be completed on the original diagnostic biopsy and the final melanoma excision
Other: Gene expression profiling — Gene expression profiling will be completed on the original diagnostic biopsy and the final melanoma excision

SUMMARY:
The purpose of this study is to determine whether a medication, fluvastatin, can change melanoma to a state that is less likely to metastasize or recur.

Fluvastatin is experimental in this setting because it is not approved by the Food and Drug Administration (FDA) for treatment or prevention of melanoma. However, fluvastatin has been approved by the FDA for treating high cholesterol.

DETAILED DESCRIPTION:
This is an open-label, single arm, study assessing the activity of fluvastatin in shifting the transcriptome in melanoma. Subjects with melanoma will be asked to participate and all subjects will receive the study drug, fluvastatin, for 2 weeks.

The primary objective of this study to determine whether administration of fluvastatin changes the melanoma transcriptome

The secondary objective of this study is to determine whether administration of fluvastatin changes the gene expression profile of Class 2 melanoma to Class 1 melanoma.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed melanoma clinically staged as AJCC Stage 1-3.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Participant having received a statin drug within 1 month of study enrollment.
* Participant receiving any other investigational agents.
* History of adverse reactions (eg. myalgias, transaminitis, or rhabdomyolysis) attributed to compounds of similar chemical or biologic composition to fluvastatin or other agents used in this study.
* Participants with uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, liver disease, or psychiatric illness/social situations that would limit compliance with study requirements.
* Participant currently pregnant (as assessed by positive pregnancy test prior to enrollment) or breastfeeding

  --Pregnant or breastfeeding women are excluded from this study because Fluvastatin has the potential for teratogenic or abortifacient effects. Women of childbearing potential will be asked to take a pregnancy test prior to enrollment (unless a pregnancy test administered within the last month is present in the medical record and is negative). A woman of childbearing potential is defined as a premenopausal female capable of becoming pregnant. Men do not need to use contraception while taking this medication.
* Participants currently receiving BRAF inhibitors, MEK inhibitors, immunotherapy, or any other non-surgical treatment for melanoma.
* Participants currently receiving nucleoside reverse transcriptase inhibitors. These participants are excluded because use of NRTIs may confound the transcriptome measurements used in this study since as described above they are predicted to modify melanoma gene expression.
* Any condition or situation that, in the investigator's opinion, may put the patient at significant risk, or may significantly interfere with the patient's participation in the study.
* Participants concurrently taking macrolide antibiotics (eg erythromycin, clarithromycin), azole antifungals (eg itraconazole, ketoconazole), protease inhibitors (eg ritonavir, telaprevir), gemfibrozil, cyclosporine, danazol, amiodarone, amlodipine, verapamil, diltiazem, azithromycin, carbamazepine, phenytoin, or rifampin are excluded.
* Participants with baseline ALT greater than 3 times the upper limit of normal.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-11-06 (Estimated); Primary Completion 2021-04-01 (Estimated); Study Completion 2021-04-01 (Estimated)

PRIMARY OUTCOMES:
Genetic profile shift in melanoma transcriptome | Two weeks
  The study team will report which of the 28 genes had significant expression changes. A 2-fold change in the appropriate direction with a p-value of at least 0.05 will be considered significant for potential therapeutic value. P-values will be corrected for the false discovery rate using the Benjamini-Hochberg procedure. Fluvastatin successful in shifting the genetic profile in a therapeutic manner if at least half of the 28 genes have significant expression changes

SECONDARY OUTCOMES:
Number of patients who convert from Class 2 to Class 1 | Two weeks
  Number of patients who convert from Class 2 to Class 1 profile on retesting

CONTACTS AND LOCATIONS:
Overall Officials: Wesley Yu, MD, Principal Investigator — University Hospitals Cleveland Medical Center, Case Comprehensive Cancer Center

IPD SHARING:
Plan to Share IPD: No
This study is a pilot study to help assess the power needed for a larger study and to determine biologic activity. If a larger study is conducted, data will be shared.